CLINICAL TRIAL: NCT07066020
Title: A Telehealth-Delivered Physical Activity Intervention Improves Sleep and Reduces Parental Stress in Children With Autism Spectrum Disorder: A Randomized Controlled Trial
Brief Title: Telehealth Exercise Boosts Sleep and Reduces Parental Stress in Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Normal University (Other)
Responsible Party: Principal Investigator, Shen Xin, Principal Investigator, Hunan Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SUS2025
Record Dates: First submitted 2025-04-24; First posted 2025-07-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder (ASD; Sleep Disturbances in Children; Parental Stress
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model in which participants (parent-child dyads) are randomized into two groups: one receiving a family-based physical activity intervention delivered via telehealth, and the other serving as a wait-list control. The intervention spans 16 weeks and includes structured online sessions, home-based exercises, and professional remote support. Outcomes will be assessed in both children and parents at multiple time points.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-Person Physical Activity (In-PA) Program (Active Comparator): Participants in this arm are assigned to a 16-week, structured, in-person physical activity regimen. Children attend three 40-minute sessions per week on-site at a partner school. Sessions are delivered by certified physical education instructors trained in a standardized protocol. The curriculum incorporates five core components: an Individualized Motor Protocol, Structured Group Sessions, Self-Management Training, Behavior Change Support, and Safety Oversight. During sessions, instructors provide hands-on correction and adjust task difficulty in real-time based on each child's motor and sensory profile. Attendance and performance are systematically recorded.
  Interventions: Behavioral: In-Person Supervised Physical Activity Program
- Telehealth-delivered Physical Activity (TPA) Program (Experimental): Participants' caregivers are assigned to a 16-week, theory-driven (Social Cognitive Theory and Self-Determination Theory) physical activity program delivered remotely. The intervention is co-facilitated by trained therapists via videoconference (Tencent VooV Meeting) in small cohorts (8-10 caregivers). The program consists of weekly 45-minute group sessions focused on personalized exercise prescription, collaborative goal setting, behavior change support, and safety education. Caregivers are instructed to guide their child through three 30-40 minute physical activity sessions per week and submit biweekly activity logs to a secure cloud platform. Based on these logs, therapists conduct two individualized 10-minute phone consultations per family during the intervention to provide tailored feedback and troubleshoot barriers. Each family receives a theory-informed workbook and supplemental materials.
  Interventions: Behavioral: Telehealth-delivered Physical Activity Program for Children with ASD
- Standard Advice and Use (SAU) (Other): Participants in this control arm receive general health promotion materials without a formal or structured physical activity prescription. At the beginning of the study, caregivers attend a one-time webinar-style group session covering general health topics, including pediatric nutrition, sleep hygiene, and caregiver stress management. Following the session, participants are provided with an exercise guidance manual authored by pediatric specialists for their optional, independent use. No structured or therapist-guided physical activity is provided, and there is no active monitoring.
  Interventions: Other: General Health Education Materials

INTERVENTIONS:
Behavioral: Telehealth-delivered Physical Activity Program for Children with ASD — This is a 16-week, theory-driven (Social Cognitive Theory & Self-Determination Theory) behavioral intervention delivered remotely to caregivers of children with ASD. The program is facilitated by trained therapists via videoconference in small groups and consists of weekly 45-minute sessions. Core components include personalized exercise prescription, collaborative goal-setting, behavior change support, and safety education. Caregivers are coached to guide their child in three 30-40 minute physical activity sessions per week. To provide individualized support, therapists conduct two 10-minute one-on-one phone consultations per family based on biweekly activity logs submitted by caregivers.
  Arms: Telehealth-delivered Physical Activity (TPA) Program
Behavioral: In-Person Supervised Physical Activity Program — This is a 16-week, structured, in-person physical activity intervention for children with ASD. The program consists of three 40-minute sessions per week delivered on-site at a partner school by certified physical education instructors. The curriculum is manualized and includes an Individualized Motor Protocol, Structured Group Sessions, and Behavior Change Support. Instructors provide direct, hands-on correction and feedback during sessions, adjusting task difficulty in real-time to match each child's individual capabilities and needs.
  Arms: In-Person Physical Activity (In-PA) Program
Other: General Health Education Materials — This is a minimal intervention control. Participants in this group do not receive a structured or guided physical activity program. At the beginning of the study, caregivers are provided with a one-time, webinar-style session on general pediatric health topics (e.g., nutrition, sleep hygiene) and an exercise guidance manual. These materials are for optional, independent use by the caregivers, and no active monitoring or follow-up is provided by the research team regarding their use.
  Arms: Standard Advice and Use (SAU)

SUMMARY:
This study aims to test whether a physical activity program delivered through telehealth can help improve sleep quality in children with autism spectrum disorder (ASD) and reduce stress and improve well-being in their parents.

Children in the study will wear a small device (an accelerometer) to measure their physical activity levels and sleep. Parents will answer questionnaires about their child's sleep habits, behavior, and social skills, as well as their own sleep, stress levels, and parenting experience.

The program will be delivered remotely, allowing families to participate from their homes. It includes guided physical activities, family-based exercises, and regular telehealth support from professionals.

The goal is to find out if this type of remote support can help both children with autism and their caregivers in daily life.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for enrollment:

The participant is a child aged 8 to 12 years with a confirmed diagnosis of Autism Spectrum Disorder (ASD) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).

A parent or primary caregiver aged 18 years or older is willing and able to participate in the study.

The child demonstrates the ability to understand and follow simple instructions necessary for study procedures.

Presence of significant parent-reported insomnia symptoms, specifically defined as having bedtime resistance, sleep-onset delay, or night awakenings that occur on five to seven nights per week, as identified using the Children's Sleep Habits Questionnaire (CSHQ).

Exclusion Criteria:

Participants will be excluded if they meet any of the following criteria:

Currently receiving, or has recently completed, pharmacological or formal behavioral treatment for sleep problems.

Presence of any medical condition that significantly limits physical activity (e.g., moderate-to-severe asthma, congenital heart disease).

Diagnosis of a complex neurological disorder (e.g., epilepsy).

Presence of other known medical or psychiatric conditions that could be the primary cause of sleep disturbance (e.g., sleep apnea, restless legs syndrome, severe anxiety).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Children's Sleep Habits Questionnaire | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  The Children's Sleep Habits Questionnaire (CSHQ) is a parent-reported tool designed to assess sleep behaviors in children aged 4 to 12. It comprises 45 items covering eight subscales: bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep-disordered breathing, and daytime sleepiness. Parents rate each item based on frequency over the past week, using a 3-point scale: "usually" (5-7 times), "sometimes" (2-4 times), or "rarely" (0-1 time). A higher total score indicates more sleep problems. The CSHQ has demonstrated good reliability and validity in identifying pediatric sleep disorders.
Objective Sleep Efficiency | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  This metric represents the percentage of time spent asleep relative to the total time a person spends in bed, calculated as (Total Sleep Time / Time in Bed) x 100. The data is objectively derived from continuous actigraphy recordings captured by a wearable accelerometer. As a primary indicator of sleep consolidation, a higher sleep efficiency percentage signifies more continuous, high-quality, and less fragmented sleep. It is a key objective marker for evaluating overall sleep quality and the effectiveness of interventions aimed at improving restorative sleep.
Objective Moderate-to-Vigorous Physical Activity | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  The average total time per day spent in physical activities of moderate-to-vigorous intensity. This outcome is objectively quantified using a wearable accelerometer and is a key indicator of health-enhancing physical activity levels.
Objective Sleep Onset Latency | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  This parameter quantifies the period of time, measured in minutes, from the designated "lights out" or the beginning of the sleep attempt, to the first epoch of consolidated sleep. This is determined through an algorithmic analysis of movement data from the wearable accelerometer, which identifies the transition from an active wakeful state to a sustained resting state. SOL is a critical objective measure of sleep initiation. A prolonged SOL is a hallmark symptom of sleep-onset insomnia, making it a valuable outcome for assessing difficulties in falling asleep.
Objective Total Sleep Duration | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  This represents the total amount of time, measured in hours, that an individual is scored as being asleep during the main nocturnal sleep period. It is distinct from "Time in Bed" because it excludes all periods of wakefulness that occur after sleep has begun (WASO). The outcome is objectively quantified using validated algorithms that analyze wrist-movement data from the accelerometer. Sufficient sleep duration is fundamental for cognitive performance, emotional regulation, and physical health, making this a critical endpoint for assessing overall sleep adequacy.
Objective Wake After Sleep Onset | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  This metric is the total duration, in minutes, of all periods of wakefulness that occur between the initial onset of sleep and the final awakening in the morning. Objectively calculated from accelerometer activity data, WASO serves as a direct biomarker of sleep fragmentation and an individual's ability to maintain sleep. Elevated WASO indicates disturbed, non-restorative sleep, which can disrupt sleep architecture and is often associated with daytime fatigue and impaired cognitive function.
Objective Number of Awakenings | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  This metric is the total count of distinct awakening episodes that are recorded after sleep has initially begun and before the final morning awakening. An algorithm identifies these events by detecting significant shifts from periods of inactivity (inferred sleep) to periods of activity (inferred wakefulness). While related to WASO, this metric specifically quantifies the frequency of sleep disruptions rather than their cumulative duration. A higher

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  Parent sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). This 19-item self-report measure generates seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of these seven component scores (each rated 0-3) creates a global PSQI score that ranges from 0 to 21, with higher scores indicating poorer sleep quality (a more negative outcome).
Hospital Anxiety and Depression Scale | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  Parental mood will be assessed using the Hospital Anxiety and Depression Scale (HADS). It contains 14 items, divided into a 7-item Anxiety subscale and a 7-item Depression subscale. Items are rated on a 4-point scale (0-3) based on the intensity or frequency of symptoms. Each subscale score ranges from 0 to 21, where higher scores indicate greater symptom severity for anxiety and depression, respectively (a more negative outcome).
Parenting Stress Scale | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  Parenting-related stress will be evaluated using the Parenting Stress Scale (PSS). This 17-item scale measures the level of stress experienced by parents by assessing both positive and negative aspects of their parenting role. Participants rate their agreement with each statement on a 5-point scale. The total score ranges from 17 to 85, with higher scores indicating a greater level of parenting stress (a more negative outcome).
Multidimensional Scale of Perceived Social Support | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  Perceived social support will be assessed using the Multidimensional Scale of Perceived Social Support (MSPSS). This 12-item scale evaluates an individual's perception of social support. Each item is rated on a 7-point scale (1 'Very Strongly Disagree' to 7 'Very Strongly Agree'). The total score ranges from 12 to 84, where higher scores indicate a greater level of perceived social support (a more positive outcome).
World Health Organization Quality of Life-BREF | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  Parental quality of life will be evaluated using the World Health Organization Quality of Life-BREF (WHOQOL-BREF). This 26-item instrument is a shorter version of the WHOQOL-100, assessing four domains: Physical Health, Psychological Health, Social Relationships, and Environment. Items are rated on a 5-point scale. For analysis, domain scores are calculated and transformed to a scale ranging from 0 to 100, where higher scores indicate a better quality of life (a more positive outcome).
Behavior Problems Inventory | Measurements will be taken at baseline (pre-intervention), after the 16-week intervention, and at 6-month and 12-month post-intervention follow-ups.
  Behavioral problems will be assessed using the Behavior Problems Inventory . This 52-item instrument evaluates challenging behaviors across three subscales: Self-Injurious Behavior, Stereotyped Behavior, and Aggressive/Destructive Behavior. Each item is rated for frequency and severity on a 4-point scale from 0 (not a problem) to 3 (a severe problem). For this study, the total BPI score, representing the sum of all 52 items, will be used for analysis. The total score ranges from 0 to 156, with higher scores indicating a greater severity of behavior problems (a more negative outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Normal University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data involving children with Autism Spectrum Disorder (ASD), individual participant data (IPD) may not be shared. This decision is based on privacy concerns, ethical considerations, and data protection regulations. Since the participants are minors, their parents have provided consent under strict confidentiality, ensuring the protection of their personal and health information.